CLINICAL TRIAL: NCT06445049
Title: Assessing Intrinsic Respiratory Rate in Mechanically Ventilated Adult Patients With Reverse Triggering as an Incentive for Accelerating Transition to Spontaneous Breathing and Extubation: Pilot Randomized Clinical Trial - INTRINSIC
Brief Title: Intrinsic Respiratory Rate Assessment During Mechanical Ventilation to Accelerate Spontaneous Breathing and Extubation
Acronym: INTRINSIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4902
Record Dates: First submitted 2024-05-30; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Reverse Triggering; Patient Ventilator Dyssynchrony
Keywords: Mechanical Ventilation; Dyssynchrony; Reverse Triggering; Intensive Care Unit
MeSH Terms: conditions — Patient-Ventilator Asynchrony

STUDY DESIGN:
Intervention Model Description: Deferred consent model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): The participant will receive the current standard intensive care.
- brief test (Active Comparator): The intervention is a simple brief test as follows: With the ventilator set with the patient clinical settings, it will be performed an up to 30sec-long or two inspiratory effort and-expiratory occlusion maneuver on the ventilator and/or switch the patient to pressure support for up to 30sec-long to assess the presence of intrinsic respiratory rate.
  If an intrinsic respiratory rate ≥8 breaths per minute is present and P/F ratio is ≥150 it will be performed a 5-minute "test" in pressure support ventilation with the pressure support level to match the clinical setting of the patient. If the patient tolerates well 5 minutes in pressure support (see criteria below) the clinical team will be informed:
  - It will be indicated that the patient tolerated 5 min of PSV and suggest to the clinicians and physician in charge to transition the patient to pressure support ventilation plus suggest reducing sedation.
  Interventions: Other: brief test

INTERVENTIONS:
Other: brief test — The intervention is a simple brief test as follows: With the ventilator set with the patient clinical settings, it will be performed an up to 30sec-long or two inspiratory effort and-expiratory occlusion maneuver on the ventilator and/or switch the patient to pressure support for up to 30sec-long to assess the presence of intrinsic respiratory rate.
  If an intrinsic respiratory rate ≥8 breaths per minute is present and P/F ratio is ≥150 it will be performed a 5-minute "test" in pressure support ventilation with the pressure support level to match the clinical setting of the patient. If the patient tolerates well 5 minutes in pressure support (see criteria below) the clinical team will be informed:
  - It will be indicated that the patient tolerated 5 min of PSV and suggest to the clinicians and physician in charge to transition the patient to pressure support ventilation plus suggest reducing sedation.
  Arms: brief test

SUMMARY:
The goal of this study is to identify patients with reverse triggering who's the potential to breath spontaneously is hidden because of the ventilator management strategy by performing a simple 30sec-test with includes reducing the support from the ventilator. The findings will provide clear advice to doctors on how to better care for these patients.

This will be a pilot randomized clinical trial including 70 adult patients (aimed at equal number of men and woman) sedated and under controlled ventilation having reverse triggering. The study will be conducted in two ICUs: 1) St. Michael's Hospital, Toronto Canada and 2) Toronto Western Hospital, Toronto, Canada.

DETAILED DESCRIPTION:
The objective of this study is to investigate the impact of assessing intrinsic respiratory rate in mechanically ventilated patients with reverse triggering on the facilitation of transition to spontaneous breathing and successful extubation.

Patients will be excluded if under current use of continuous neuromuscular blocking agent or severe metabolic acidosis (Ph<7.25 at the time of study procedure.

Patients will be screened every morning from 8:00 am to 9:00 am all the patients under controlled ventilation to detect the presence of reverse triggering by looking at the screen on the ventilator (2-5 min observation). The research team (research MDs, physiotherapists and respiratory therapists) is very well trained at detecting reverse triggering. Patients will then be randomized to standard of care or intervention using a deferred consent model.

* Control group: standard care.
* Intervention group: The intervention is a simple brief test as follows: With the ventilator set with the patient clinical settings, it will be performed an up to 30sec-long or two inspiratory effort and expiratory occlusion maneuver on the ventilator and/or switch the patient to pressure support for up to 30sec-long to assess the presence of intrinsic respiratory rate.

If an intrinsic respiratory rate ≥8 breaths per minute is present and P/F ratio is ≥150 it will be performed a 5-minute "test" in pressure support ventilation with the pressure support level to match the clinical setting of the patient. If the patient tolerates well 5 minutes in pressure support (see criteria below) the clinical team will be informed:

- It will be indicated that the patient tolerated 5 min of pressure support ventilation and suggest to the clinicians and physician in charge to transition the patient to pressure support ventilation plus suggest reducing sedation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aimed at equal number of men and woman) sedated and under controlled ventilation having reverse triggering.

Exclusion Criteria:

* under current use of continuous neuromuscular blocking agent or severe metabolic acidosis (Ph<7.25) at the time of study procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients tolerating the transition to assisted breathing, or having an SBT, or being extubated within 48 hours | 48 hours
  Number of patients tolerating the transition to assisted breathing (e.g., Pressure Support Ventilation, Neurally Adjusted Ventilatory Assist, Proportional assist ventilation with load-adjustable gain factors), or having an SBT, or being extubated within 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Brochard, Principal Investigator — Unity Health Toronto - St. Michael's Hospital

REFERENCES:
- [Background] Rodrigues A, Telias I, Damiani LF, Brochard L. Reverse Triggering during Controlled Ventilation: From Physiology to Clinical Management. Am J Respir Crit Care Med. 2023 Mar 1;207(5):533-543. doi: 10.1164/rccm.202208-1477CI. PMID 36470240